CLINICAL TRIAL: NCT06692556
Title: Randomized Comparative Multicenter Phase III Study of a Strategy Integrating Adjuvant Radiation Therapy Versus Strategy Based on Monitoring in the Treatment of Carcinomas Spinocellular With High Risk of Recurrence
Brief Title: Study of a Strategy Integrating Adjuvant Radiation Therapy Versus Strategy Based on Monitoring in the Treatment of Carcinomas Spinocellular With High Risk of Recurrence
Acronym: SPINO-RT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPINO-RT (ET24-046)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Squamous Cell Carcinoma (CSCC)
Keywords: Squamous cell carcinomas at high risk of recurrence; Adjuvant radiotherapy; Surveillance; Peri Nervous System Sheathing
MeSH Terms: interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized (ratio 1:1) using an online platform into one of the two study arms:
  * "Adjuvant radiotherapy" arm (=133),
  * "Surveillance" arm (n=133)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant radiotherapy (Active Comparator): Radiation therapy should be started within 8 to 10 weeks after surgery.
  An equivalent dose of 45 to 50 Gy will be delivered on the operating bed. The irradiation techniques used may be either external radiation therapy with high-energy photons or electrons or brachytherapy. Patients will be monitored regularly until the date of the first local, regional or metastatic relapse, or until the date of death if they do not relapse.
  Regardless of the type of relapse, remedial treatments will be left to the The investigator's discretion; they will be collected in the data collection book as well as data on subsequent relapses, up to the first metastatic relapse.
  Interventions: Radiation: Adjuvant radiotherapy
- Surveillance (No Intervention): Patients will not receive any treatment after surgery and will be monitored regularly until the date of their first local, regional or metastatic relapse, or until the date of death if they do not relapse.
  Regardless of the type of relapse, the treatment to be used is left to the discretion of the investigator; it will be collected in the data collection book as well as data on subsequent relapses up to the first metastatic relapse.

INTERVENTIONS:
Radiation: Adjuvant radiotherapy — Patients will receive an adjuvant radiotherapy corresponding to an equivalent dose of 45 to 50 Gy (Equivalent Dose in 2 Gy Fractions [EQD2] with a tumor alpha/beta ratio of 10 Gy) delivered on the operating bed.
  Patients will be treated by :
  * either external radiation therapy using high-energy electrons or photons:
    * 45 Gy in 15 fractions of 3 Gy
    * 50 Gy in 25 fractions of 2 Gy
  * or interstitial brachytherapy or brachytherapy via skin applicators:
    * 36 Gy in 8 fractions of 4.5 Gy
    * 36 Gy in 9 fractions of 4 Gy
    * 40 Gy in 8 fractions of 5 Gy
  Radiation therapy should be started within 8 weeks after surgery (or 10 if delayed healing).
  Patients will be monitored regularly until the date of the first relapse (local, regional or metastatic), or until the date of death (if no relapse).
  Regardless of the type of relapse, remedial treatments will be left to the the investigator's discretion up to the first metastatic relapse.
  Arms: Adjuvant radiotherapy

SUMMARY:
The goal of this clinical trial is to evaluate a strategy integrating adjuvant radiation therapy versus strategy based on monitoring in the treatment of carcinomas spinocellular with high risk of recurrence (SCC).

The investigators will compare the disease-free survival (DFS) of patients treated with adjuvant radiation therapy versus surveillance in high risk of recurrence SCC.

The main question it aims to answer is:

Is DFS different between the "adjuvant radiotherapy" group and the "surveillance" group?

Participants will:

* be distributed in one of the two arms
* will be followed up every 4 months for 2 years, then every 6 months (clinical examination, identification of concomitant treatments, imaging, quality-of-life questionnaire)
* followed up until their death or their progression whether local, regional or metastatic

DETAILED DESCRIPTION:
The use of adjuvant radiotherapy appears to provide clinical benefit, both theoretically and based on available retrospective data. This is why some patients already benefit from this complementary treatment. However, given the lack of prospective data, the use of adjuvant radiotherapy is based on heterogeneous criteria, depending on the choice of the clinician in charge of the patient or the habits of his institution.

The sponsor team therefore propose to conduct a national prospective study to compare the efficacy and safety of a strategy integrating adjuvant radiotherapy versus a strategy based on surveillance in patients with SCC at high risk of recurrence.

Considering that there is no validated standard after surgery for patients with a high risk of recurrence, it is not possible to determine a standard arm and an experimental arm. This study therefore falls within the framework of a Research Involving the Human Person of Category 2.

This protocol constitutes the first prospective evaluation of adjuvant radiotherapy, within the framework of a comparative study. This study will thus make it possible to avoid the use of this therapeutic alternative, without rigorous evaluation in a prospective framework. Its robust methodology will make it possible to determine whether adjuvant radiotherapy provides a clinical benefit to patients at high risk of recurrence. It will modify the standards of care for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age at the time of signing informed consent to participate;
* Patient with histologically confirmed, localized skin squamous cell carcinoma; Note bene: patients with carcinoma of the external auditory canal may be included in the study;
* Patient treated with complete excision surgery (R0), regardless of margin (inframillimetric or supramillimetric);
* High risk disease defined by: presence of a microscopic PNI without/with another risk factor (among those mentioned below) OR presence of 2-3 risk factors other than microscopic PNI; Note Bene: The risk factors selected are immunosuppression (only haematopathy with or without treatment) , a tumor diameter >20mm, specific location (lip/ear/temple), deep invasion (thickness >6mm or invasion beyond subcutaneous fat), low differentiation or desmoplasia;
* Patient informed and having signed consent to participate in the study;
* Patient affiliated with a health insurance plan (or beneficiary of such a plan).

Exclusion Criteria:

* Patient with in situ or mixed SCC;
* History of SCC at high risk of relapse in the same territory (head and neck, trunk or limb) in the 2 years preceding the date of randomization;
* History of SCC having received systemic treatment;
* Patient with SCC located in the endonasal, intra-oral, anogenital or vulvar mucosa;
* Patient with recurrent SCC or SCC at very high risk of relapse defined by one of the following criteria:

  * PNI with > 2 other risk factors,
  * > 3 risk factors,
  * bone invasion,
  * immunosuppression by immunosuppressive treatments (whatever the reason).
* Patient with SCC with a single risk factor other than PNI;
* Patient with SCC with lymph node or distant metastasis;
* Patient with a history of solid cancer undergoing chemotherapy;
* Patient with a contraindication to radiotherapy;
* Patient with a history of radiotherapy in the area of the lesion;
* Participation in another clinical trial that may interfere with the assessment of the primary endpoint;
* Patient under guardianship or curatorship or deprived of liberty;
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Up to 54 months
  DFS is defined as the time from the date of randomization to the date of recurrence (local, lymph node or metastatic) or death from any cause. A new skin lesion will not be considered a statistical event. Patients without an event at the date of analysis will be censored at the last date of new disease-free status.
  DFS will be estimated by the Kaplan Meier method and described in terms of median in each arm. DFS distributions will be compared between arms using a Log-Rank test. The hazard ratio from a Cox model will be calculated and presented with its 95% confidence interval. The rate of patients without recurrence at 1 and 2 years post-randomization will also be presented with their associated confidence interval.

SECONDARY OUTCOMES:
Local recurrence-free survival (lrFS) | Up to 54 months
  lrFS is defined as the time elapsed between the date of randomization and the date of metastatic recurrence or death from any cause. Patients without events at the analysis date will be censored at the last date of news without local disease. Death or metastatic recurrence will be considered as competing events.
Metastatic recurrence-free survival (mFS) | Up to 54 months
  mFS is defined as the time elapsed between the date of randomization and the date of metastatic recurrence or death from any cause. Patients without an event at the analysis date will be censored at the last date of news without metastatic disease.
Overall Survival (OS) | Up to 54 months
  OS is defined as the time from the date of randomization to the date of death from any cause. Patients without an event at the analysis date will be censored at the last date of death-free news.
Tolerance/toxicity | Up to 54 months
  The safety will be described according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTC AE) Version 5 grid by reporting the number and percentage of patients with toxicity by grade. Adverse events will be coded according to the MedDRA® dictionary and will be described by System Organ Class and Preferred Term. The number of patients with at least one AE by grade, at least one AE related to treatment, at least one serious AE (according to pharmacovigilance), at least one serious AE related to treatment will be described by treatment arm. A listing of serious AEs will be published
Quality of Life (QoL) | Up to 54 months
  QoL, will be assessed using the EORTC QLQ-C30 and the EORTC QLQ-ELD14 for the patients ≥ 75 years of age. The difference between the scores at inclusion and during follow-up will be calculated per patient. A difference of 10 points on each score will be considered clinically relevant. A graphic representation in the form of a spider plot will allow to globally visualize the evolution on all the items between the different measurement times.
Interest of radiotherapy in the subgroup of patients over 75 years old | Up to 54 months
  Due to the stratification, the aged population will be well distributed in a balanced way between the treatment arms. The main efficacy criterion and quality of life of this subpopulation will be studied in more detail.
Interest of radiotherapy in the subgroup of patients with Perineural Neoplastic Invasion (PNI) | Up to 54 months
  Due to the stratification, the population with PNI will be well balanced among the treatment arms. The main efficacy criterion and quality of life of this subpopulation will be studied in more detail.

OTHER OUTCOMES:
Progression-free survival after local recurrence salvage therapy in the Surveillance group | Up to 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Mona AMINI-ADLE, Dr, Principal Investigator — Centre Leon Berard
Locations (22):
- France (22):
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Centre Hospitalier Romans - Hopitaux Drôme Nord, Romans-sur-Isère, Drôme
  - Centre de Radiothérapie Marie Curie, Valence, Drôme
  - Centre Hospitalier de Valence, Valence, Drôme
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan, Brest, Finistère
  - Centre Hospitalier Universitaire de Bordeaux, Pessac, Gironde
  - Centre Hospitalier Annecy Genevois, Épagny-Metz-Tessy, Haute-Savoie
  - Centre Hospitalier Universitaire de Rennes, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire de Grenoble-Alpes, La Tronche, Isère
  - Centre Hospitalier Simone Veil de Blois, Blois, Loir-et-Cher
  - Centre Hospitalier Universitaire de Nantes - Hôtel-Dieu, Nantes, Loire-Atlantique
  - Institut Godinot, Reims, Marne
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, MMeurthe-et-Moselle
  - Groupe Hospitalier Bretagne Sud, Lorient, Morbihan
  - Centre hospitalier de Roanne, Roanne, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Saint-Etienne - Hôpital Nord, Saint Priest En Jarez, Pays de la Loire Region
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Puy-de-Dôme
  - Centre Hospitalier Universitaire Rouen - Hôpital Charles Nicolle, Rouen, Seine-Maritime
  - Centre Hospitalier Universitaire Amiens-Picardie, Amiens, Somme
  - Hôpital d'instruction des armées Sainte-Anne, Toulon, Var
  - Centre Léon Bérard, Lyon
  - Hôpital Bichat Claude-Bernard, Paris, Île-de-France Region